CLINICAL TRIAL: NCT01693289
Title: Phase 1 Study of Efficacy of Combined Metformin-letrozole in Comparison With Bilateral Ovarian Drilling in Clomiphene-resistant Infertile Women With Polycystic Ovarian Syndrome
Brief Title: Study to Compare Between Combimed Metformin-letrozole and Ovarian Drilling in Pcos With Bilateral Ovarian Drilling in Clomiphene-resistant Infertile Women With Polycystic Ovarian Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, IBRAHIM ABD ELGAFOR, obstetrics and gynecology department, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: elsharkwy t
Record Dates: First submitted 2012-09-23; First posted 2012-09-26 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Focus of Study
Keywords: Metformin; letrozole; ovarian drilling; clomiphene resistance; polycystic ovary.
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Letrozole

ARMS (2):
- Metformin plus letrozole (Experimental): metformin :850mg tablets twice daily for 6 months letrozole :5mg tablets twice daily form day 3to7 of cycle
  Interventions: Drug: metformin plus letrozole
- ovarian drilling (Experimental): bilateral diathermy ovarian drilling, four drills each ovary
  Interventions: Procedure: ovarian drilling

INTERVENTIONS:
Drug: metformin plus letrozole
  Other Names: cidophage plus fumara
  Arms: Metformin plus letrozole
Procedure: ovarian drilling
  Other Names: ovarian dithermy drilling
  Arms: ovarian drilling

SUMMARY:
the study compare the hormonal-metabolic and reproductive outcome between combined metformin-letrozole and ovarian drilling in clomiphene resistant women with polycystic syndrome

ELIGIBILITY:
Inclusion Criteria:

* polycystic ovary syndrome
* infertility
* clomiphene citrate resistance

Exclusion Criteria:

* women with other causes of infertility as male factor or tubal factor, those with endocrine disorders as thyroid dysfunction and hyperprolactinemia women who received hormonal treatment or ovulation induction drugs 3 months prior to the study
* pregnancy during follow up

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
hormonal and metabolic changes | 6 months

SECONDARY OUTCOMES:
reproductive outcome | 6months

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Egypt